CLINICAL TRIAL: NCT02640352
Title: A Randomized, Double Blind, Placebo-controlled Study to Investigate the Effect of a Probiotic Product on Acute Upper Respiratory Tract Infections (Common Cold) in Healthy Children
Brief Title: The Efficacy of a Probiotic Product on Acute Upper Respiratory Tract Infections (Common Cold) in Healthy Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probi AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PROIMKID_15
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Acute Upper Respiratory Tract Infections (Common Cold)
MeSH Terms: conditions — Common Cold

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probi Defendum (Active Comparator): Dietary supplement (tablet) with probiotics
  Interventions: Dietary Supplement: Probi Defendum
- Placebo (Placebo Comparator): Dietary supplement (tablet) without probiotics
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probi Defendum
  Arms: Probi Defendum
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
The aim of the present study is to test the efficacy of the combination of two probiotic bacteria in reducing the severity of upper respiratory tract infections (common cold) in healthy children attending day care or school. The probiotic bacteria used are Lactobacillus plantarum strain DSM 15312 and Lactobacillus paracasei DSM 13434 at a total dose of 1 x 10^9 CFU/tablet and day and will be consumed for a period of 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Parents / legal guardians signed written informed consent to participate in the study.
2. Healthy children (male and female) aged 3 to 7 years old (inclusive) at enrollment.
3. Children attending day care center or school.
4. No consumption of commercial products containing probiotics during the whole study period.
5. Children not being intensive consumers of regular yoghurts (no more than one 125 g serving per day).
6. Ability of the parents / legal guardians (in the Investigator's opinion) to comprehend the full nature and purpose of the study.
7. Parents' / legal guardians' consent to the study and willing to comply with all its procedures.

Exclusion Criteria:

Children presenting one or more of the following criteria will not be eligible to enter the study.

1. Flu vaccine administration within the last 3 months prior to enrollment.
2. Use of antibiotics within the last 30 days prior to enrollment.
3. Acute infection or fever at enrollment.
4. Any congenital or chronic disease that in the opinion of the investigator would adversely affect the results of the study.
5. Any kind of immunodeficiency or allergy (including known food allergy).
6. Subjects with known hypersensitivity or allergy to any component of the study products.
7. Significant illness within the 2 weeks prior to the enrollment or any active systemic infection or medical condition that may require treatment or therapeutic intervention during the study.
8. Currently participating or having participated in another clinical trial during the last 4 weeks prior to the beginning of this study.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 550 (Actual)
Dates: Start 2015-12; Primary Completion 2017-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Severity of acute upper respiratory tract infections (common cold), by means of the validated Canadian Acute Respiratory Illness and Flu Scale (CARIFS) questionnaire (total sum score), during 12 weeks of daily intake of either Probi Defendum® or placebo. | 12 weeks

SECONDARY OUTCOMES:
Number of common cold episodes | 12 weeks
Duration of common cold episodes | 12 weeks
Incidence of common cold episodes | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- AO L. Sacco, Milan, Italy

IPD SHARING:
Plan to Share IPD: No